CLINICAL TRIAL: NCT06751719
Title: Combined Effects of Proprioceptive, Calisthenic, and Kinesthetic Exercises on Pain, Range of Motion, and Functional Disability in Chronic Low Back Pain
Brief Title: Proprioceptive, Calisthenic, and Kinesthetic Exercises for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hatoma Fatima Malik
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: Chronic Low Back Pain; Calisthenic exercises; Proprioceptive exercises; Kinesthetic exercises; Disability
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): This control group will only participate in core stabilization exercises and heat therapy. The exercise session would be held 3 times a week.
  Interventions: Other: core stabilization exercises; Other: heat therapy
- Group B (Experimental): This intervention group will consist of participants who will engage in proprioceptive, calisthenic, and kinesthetic exercises along with core stabilization exercises and heat therapy. The exercise session would be held 3 times a week.
  Interventions: Other: core stabilization exercises; Other: heat therapy; Other: proprioceptive exercises; Other: calisthenic exercises; Other: kinesthetic exercises

INTERVENTIONS:
Other: core stabilization exercises — The core exercises would be held for 7 to 8 seconds, repeated 10 times, and rest for 3 seconds between repetitions and 1 minute rest between each exercise. These exercises will include:
  1. Abdominal hollowing
  2. Supine extension bridge
  3. Partial Curls
Other: heat therapy — The heat therapy would be applied to the lumbar region for 10 minutes.
Other: proprioceptive exercises — The proprioceptive exercises will include rest for 3 seconds between repetitions and 1-minute rest between each exercise. These exercises will include:
  1. One leg balance - 10 seconds hold time with 3 repetitions
  2. Forward leg swings - 15 swings
  3. Sideways leg swings - 15 swings
  Arms: Group B
Other: calisthenic exercises — The calisthenic exercises will include:
  1. Abductor's leg raise for 10 repetitions
  2. Prone leg extension for 10 repetitions
  3. Alternate toe touch for 10 repetitions
  Arms: Group B
Other: kinesthetic exercises — The kinesthetic exercises will have 1 minute rest in between exercises. These exercises will include:
  1. Toe walking for 20 meters distance
  2. Heel walking for 20 meters distance
  Arms: Group B

SUMMARY:
Numerous studies have emphasized the debilitating effects of chronic low back pain (CLBP), which persists for over 12 weeks and impacts approximately 20% of the global population. The etiology of CLBP encompasses various factors, such as sedentary lifestyles, diminished muscle strength, poor neuromuscular control of deep trunk muscles, and compromised proprioception, all contributing to lumbar spine strain. These factors result in limitations in essential daily activities, significantly diminishing the overall quality of life. Continued exploration in this field is essential to furthering our understanding of managing chronic low back pain. Investigating alternative treatment approaches, such as proprioceptive, calisthenic, and kinesthetic exercises, contributes to expanding the range of solutions available for addressing this issue. Embracing a diverse array of interventions not only proves beneficial but also holds promise in providing long-term advantages for enhancing patients' overall well-being. Therefore, this study aims to comprehensively investigate the combined effects of proprioceptive, kinesthetic, and calisthenic exercises, alongside core stabilization exercises, in alleviating chronic low back pain and their potential to enhance range of motion and diminish functional disability in individuals with CLBP in Lahore, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 3 months or above LBP
* Moderate pain (NPRS: 3-7)
* Disability score of 19% or greater as evident from the modified Oswestry Disability Questionnaire (MODQ)

Exclusion Criteria:

* History of inflammatory joint diseases e.g. rheumatoid arthritis, gouty arthritis, psoriatic arthritis, and ankylosing spondylitis
* History of neurological deficit e.g. paresthesia, sensory loss, radiculopathy, myelopathy
* History of surgery related to spine, lower extremities, metal implants on lower extremities
* History of any mental illness
* Subjects on medication e.g. antidepressants, corticosteroids, and anti-inflammatory medications
* Other conditions include peripheral vascular diseases, recent fractures including lower limb or spine, osteoporosis, spine or other joint deformities, brain injuries, neuromuscular disorders, and respiratory diseases
* Pregnancy

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
numeric pain rating scale (NPRS) | baseline, after 4 weeks
  A numeric pain rating scale (NPRS) would be used to assess the patient's pain measure for chronic low back pain before and after exercises. This 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). The NPRS has a validity of 0.86 to 0.95 and a reliability of 0.96.
inclinometer | baseline, after 4 weeks
  An inclinometer would be used to measure the range of motion for the lumbar spine. The inclinometer for lumbar ROM has a reliability of 0.97.
Modified ODI for disability (Urdu version) | baseline, after 4 weeks
  Modified ODI for disability (Urdu version) would be used to assess the patient's functional disability for chronic low back pain at 0 weeks and then at 4 weeks. The modified ODI has a reliability of 0.90. For each question, 0 points is the minimum, and 5 points is the maximum. Add up the total score for 10 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Study Director — Riphah International University, Lahore; Hatoma Fatima Malik, DPT, Principal Investigator — Riphah International University, Lahore
Locations (1):
- Riphah Rehab Training and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No